CLINICAL TRIAL: NCT02255968
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Multiple-Dose Safety, Tolerability, and Pharmacokinetic Study of EDP-788 in Healthy Adult Volunteers
Brief Title: Evaluation of the Safety, Tolerability, and Pharmacokinetics of Multiple Oral Doses of EDP-788
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EDP788-002
Record Dates: First submitted 2014-07-29; First posted 2014-10-03 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Normal Volunteers; Safety; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EDP-788 (Experimental): Multiple doses with dose escalation to continue in successive cohorts
  Interventions: Drug: EDP-788
- Placebo (Placebo Comparator): Multiple doses with dose escalation to continue in successive cohorts
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-788 — EDP-788 Capsules. All interventions are given as multiple doses.
  Arms: EDP-788
Drug: Placebo — Matching placebo capsules. All interventions are given as multiple doses
  Arms: Placebo

SUMMARY:
The primary objective of the study is to determine the safety and tolerability of multiple doses of orally administered EDP-788. Secondary objectives of the study are to describe the pharmacokinetics of EDP-788 (and its metabolite EDP-322) after multiple doses of orally administered drug.

DETAILED DESCRIPTION:
Three cohorts of subjects will be enrolled to receive either EDP-788 or placebo. The dose of EDP-788 will be increased with each successive cohort. In addition, a 4th cohort may be enrolled, depending on clinical findings (tolerability, safety, pharmacokinetics) observed in the first 3 cohorts. In each cohort, 8 subjects will receive a q12h oral dose regimen of EDP-788 (6 subjects) or placebo (2 subjects). All subjects receive multiple doses of study drug (EDP-788 or placebo).

ELIGIBILITY:
Key Inclusion Criteria:

* In good general health
* BMI between 18 - 32 kg/m2
* Women must be of non-childbearing potential (surgically sterilized)
* Normal electrocardiogram
* Willing to abstain from strenuous physical exercise starting 3 days prior to admission to the study clinic through the 17 - 19 day post-dosing visit

Key Exclusion Criteria:

* Hypersensitivity to macrolide antibiotics
* Abnormal laboratory values
* Gastroenteritis within 1 week of study drug administration
* Use of any investigational drugs within 28 days of study drug administration
* History of gastrointestinal surgery which may interfere with drug absorption
* Active Hepatitis B, Hepatitis C, or HIV infection
* Use of prescription or non-prescription drugs within 14 days of study drug administration
* Use of nicotine within 3 months of study drug administration

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | From time of dosing to 20-23 days after receiving last dose of study drug

SECONDARY OUTCOMES:
Changes from baseline in laboratory values and vital signs | From time of dosing to 20-23 days after receiving last dose of study drug
Pharmacokinetic parameters | From time of dosing to 3 days after receiving the last dose of study drug
  As measured by peak plasma concentration (Cmax)

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Phase 1 Clinic, Austin, Texas, United States